CLINICAL TRIAL: NCT05654324
Title: Investigation of Acute Effect of Pelvic Floor Muscle Exercises on Inferior Vena Cava
Brief Title: The Effect of Pelvic Floor Muscle Exercises on the Inferior Vena Cava
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir University of Economics (Other)
Responsible Party: Principal Investigator, Seda Yakit Yesilyurt, Lecturer Dr, Izmir University of Economics
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: İEÜ_SYY
Record Dates: First submitted 2022-11-30; First posted 2022-12-16 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Supine Hypotensive Syndrome

STUDY DESIGN:
Intervention Model Description: This research is a prospective and controlled study. The data of the study will be collected from pregnant women (Experimental group) and non-pregnant women (Control group).
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregnant women (Experimental): Pregnant women aged 18-40, 20-40 weeks of gestation.
  Interventions: Other: pelvic floor muscle exercises
- Non-Pregnant (Active Comparator): Being a non-pregnant woman who is in the same age range as the experimental group.
  Interventions: Other: pelvic floor muscle exercises

INTERVENTIONS:
Other: pelvic floor muscle exercises — Before the pelvic floor exercises are taught to all women participating in the study, a brief informational training about the function and structure of the pelvic floor and pelvis will be given using visuals. The application protocol will be given by experienced specialist physiotherapists who have received special training on pelvic floor muscle training. In this study, the training protocol described by Mørkved et al and Bø et al will be used. An exercise series will consist of slow and fast muscle contractions of the pelvic floor muscles. The exercise series will include 10 reps of maximum pelvic floor muscle contraction held for 6 seconds followed by three rapid muscle contractions. A 10-second rest period will be given between each exercise series. A total of 5 minutes, 4 repetitions of pelvic floor muscle contraction series will be applied, including the rest period.

SUMMARY:
The aim of this study is to examine the effect of pelvic floor muscle exercises on the hemodynamic responses of the vena cava inferior in pregnant and non-pregnant women.

DETAILED DESCRIPTION:
The IVC is responsible for approximately two-thirds of the total venous return to the heart. The blood flow in the IVC is affected by the respiratory and cardiac cycle. One of the factors affecting blood flow is pregnancy. Studies have shown that the hemodynamic responses of the IVC may vary depending on the position, and that the supine position puts pressure on the IVC during pregnancy.

Compression of the growing fetus against the IVC can cause supine hypotensive syndrome and fetal danger. However, there is no definite finding about the effects of exercise performed in the supine position. Jefferys et al. reported that the reduction in blood flow at rest is twice that that occurs during exercise and that the level of blood flow should not be a cause for concern in healthy asymptomatic women who choose to exercise in the supine position in late pregnancy. Based on this information, we predict that pelvic floor muscle exercises can change the hemodynamic responses of the IVC and reduce the compression on it.

In order to evaluate the effect of pelvic floor muscle exercises on hemodynamic responses of IVC and compression on it, pregnant and non-pregnant women will be measured by ultrasonography. Women eligible for the study will be seated and rested for 30 minutes before taking the measurement. Then, he will be taken to the supine position, rested for 2 minutes, and the first measurements will be taken at the 3rd minute. pelvic floor muscle exercises will be applied for 5 minutes as stated in the literature. Ultrasonographic measurements will be repeated in the supine position immediately after the pelvic floor exercises and 5 minutes after the exercise. Measurements will be applied to all participants in the same order. During the exercises blood pressure, heart rate and peripheral oxygen saturation will be monitored. Before and after the exercises, the heart rate and blood pressure parameters of the women will be recorded.

ELIGIBILITY:
Inclusion Criteria:

Experimental group

* Being pregnant between the ages of 18-40,
* At least primary school graduate and able to read and write,
* The gestational age is 20-40 weeks,
* Not having any mental problems that prevent cooperation and understanding.

Control group

* Being a non-pregnant woman who is in the same age range as the experimental group,
* At least primary school graduate and able to read and write,
* Not having any mental problems that prevent cooperation and understanding.

Exclusion Criteria:

* Pregnant women with acute or chronic diseases with poor placental adaptation and vascular damage such as diabetes, chronic arterial hypertension and preeclampsia, as the fetus is closer to the threshold of hypoxia and acidemia and adaptive phenomena may fail,
* Pregnant women with intra-uterine growth restriction and fetal anomaly,
* Pregnant women with cardiovascular disease,
* Pregnant women considered as high risk by the obstetrician,
* Pregnant women with premature, premature birth or miscarriage risk,
* Pregnant women diagnosed with neurological disease,
* Obese women (body mass index > 30),
* Women whose IVC measurements cannot be made with ultrasonography,
* Women with severe low back pain (not able to do housework regularly),
* Women who have been diagnosed with a psychiatric illness,
* Women with a history of gynecological surgery,
* Women with pelvic floor dysfunction,
* Women who cannot lie in the supine position.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Change of the collapsibility index (%) of IVC | immediately after the intervention
  The collapsibility index (%) of IVC will be calculated using the formula:
  [(Maximum IVC diameter - Minimum IVC diameter)/Maximum IVC diameter] × 100.
Change of Pulsatility index of IVC | immediately after the intervention
  Doppler (Toshiba Medical Systems, Aplio 400, Berlin) flow velocimetry will be evaluated.
Changes of IVC diameters | immediately after the intervention
  M mode ultrasonography will be used for expiratory (IVC d min) and end-inspiratory (IVC d min) diameter measurement.

SECONDARY OUTCOMES:
Change of the collapsibility index (%) of IVC | 5 minutes after the intervention
  The collapsibility index (%) of IVC will be calculated using the formula:
  [(Maximum IVC diameter - Minimum IVC diameter)/Maximum IVC diameter] × 100.
Change of Pulsatility index of IVC | 5 minutes after the intervention
  Doppler (Toshiba Medical Systems, Aplio 400, Berlin) flow velocimetry will be evaluated.
Changes of IVC diameters | 5 minutes after the intervention
  M mode ultrasonography will be used for expiratory (IVC d min) and end-inspiratory (IVC d min) diameter measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University İzmir Tepecik Education and Research Hospital Gynecology and Obstetrics Clinic, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klein-Weigel PF, Elitok S, Ruttloff A, Reinhold S, Nielitz J, Steindl J, Lutfi P, Rehmenklau-Bremer L, Hillner B, Fuchs H, Wrase C, Herold T, Beyer L. Inferior vena cava-syndrome. Vasa. 2021 Jul;50(4):250-264. doi: 10.1024/0301-1526/a000919. Epub 2021 Jan 18. PMID 33459041
- [Background] Gagne MP, Richebe P, Loubert C, Drolet P, Gobert Q, Denault A, Zaphiratos V. Ultrasound evaluation of inferior vena cava compression in tilted and supine term parturients. Can J Anaesth. 2021 Oct;68(10):1507-1513. doi: 10.1007/s12630-021-02051-w. Epub 2021 Jul 1. PMID 34212308
- [Background] Fields JM, Catallo K, Au AK, Rotte M, Leventhal D, Weiner S, Ku BS. Resuscitation of the pregnant patient: What is the effect of patient positioning on inferior vena cava diameter? Resuscitation. 2013 Mar;84(3):304-8. doi: 10.1016/j.resuscitation.2012.11.011. Epub 2012 Nov 21. PMID 23178869
- [Background] Practice Guidelines for Obstetric Anesthesia: An Updated Report by the American Society of Anesthesiologists Task Force on Obstetric Anesthesia and the Society for Obstetric Anesthesia and Perinatology. Anesthesiology. 2016 Feb;124(2):270-300. doi: 10.1097/ALN.0000000000000935. No abstract available. PMID 26580836
- [Background] Supine lying during pregnancy. Journal of Pelvic, Obstetric and Gynaecological Physiotherapy. 2018; 122:77-83
- [Background] Jeffreys RM, Stepanchak W, Lopez B, Hardis J, Clapp JF 3rd. Uterine blood flow during supine rest and exercise after 28 weeks of gestation. BJOG. 2006 Nov;113(11):1239-47. doi: 10.1111/j.1471-0528.2006.01056.x. Epub 2006 Sep 15. PMID 16978230
- [Background] Kim DR, Wang E. Prevention of supine hypotensive syndrome in pregnant women treated with transcranial magnetic stimulation. Psychiatry Res. 2014 Aug 15;218(1-2):247-8. doi: 10.1016/j.psychres.2014.04.001. Epub 2014 Apr 12. PMID 24768354
- [Background] Finnerty NM, Panchal AR, Boulger C, Vira A, Bischof JJ, Amick C, Way DP, Bahner DP. Inferior Vena Cava Measurement with Ultrasound: What Is the Best View and Best Mode? West J Emerg Med. 2017 Apr;18(3):496-501. doi: 10.5811/westjem.2016.12.32489. Epub 2017 Feb 24. PMID 28435502
- [Background] Shailja S, Gupta I, Suri V. Inferior vena cava diameters in pregnant women for prediction of pregnancy-induced hypertension. Int J Gynaecol Obstet. 2004 Feb;84(2):164-5. doi: 10.1016/S0020-7292(03)00157-7. No abstract available. PMID 14871520
- [Background] Singh Y, Anand RK, Gupta S, Chowdhury SR, Maitra S, Baidya DK, Singh AK. Role of IVC collapsibility index to predict post spinal hypotension in pregnant women undergoing caesarean section. An observational trial. Saudi J Anaesth. 2019 Oct-Dec;13(4):312-317. doi: 10.4103/sja.SJA_27_19. PMID 31572075
- [Background] Dodhy AA. Inferior Vena Cava Collapsibility Index and Central Venous Pressure for Fluid Assessment in the Critically Ill Patient. J Coll Physicians Surg Pak. 2021 Nov;31(11):1273-1277. doi: 10.29271/jcpsp.2021.11.1273. PMID 34689482
- [Background] Morkved S, Bo K, Schei B, Salvesen KA. Pelvic floor muscle training during pregnancy to prevent urinary incontinence: a single-blind randomized controlled trial. Obstet Gynecol. 2003 Feb;101(2):313-9. doi: 10.1016/s0029-7844(02)02711-4. PMID 12576255